CLINICAL TRIAL: NCT07316842
Title: Prospective, Single-cohort, Observational Clinical Study Evaluating the Rate of Achieving SVR12 in Patients With Chronic Hepatitis C Genotype 3 With Fibrosis Stage F0-F2 Who Received Ravidasvir + Sofosbuvir Therapy.
Brief Title: SVR12 in Genotype 3 HCV (F0-F2) Treated With RDV + SOF
Status: Active, not recruiting | Type: Observational
Sponsor: Center of target therapy (Other)
Responsible Party: Sponsor
Other Study IDs: CTT-004
Record Dates: First submitted 2025-12-01; First posted 2026-01-05 (Actual); Last update posted 2026-01-05 (Actual); Status verified 2025-12

CONDITIONS: Viral Hepatitis C
Keywords: Ravidasvir; Sofosbuvir
MeSH Terms: conditions — Hepatitis C

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study will follow a group of people with chronic hepatitis C infection of genotype 3 who have mild to moderate liver fibrosis (stages F0-F2, measured by a liver stiffness test). All participants will be receiving the antiviral drugs ravidasvir and sofosbuvir as part of their regular medical care.

Only patients who start this treatment, meet the study's eligibility criteria, and give written consent for their medical data to be used in research will take part. They will be monitored during their routine clinic visits while receiving the two-drug therapy.

After 8 weeks of treatment, researchers will check how many patients have cleared the virus from their blood. Those who achieve this response will continue to be followed for another 4 and 12 weeks after treatment to see if the virus remains undetectable.

DETAILED DESCRIPTION:
An observational, prospective, single-cohort study will be conducted in patients with chronic hepatitis C virus infection of genotype 3 and fibrosis stage F0-F2 according to the METAVIR score based on liver elastography data, who have initiated antiviral therapy with ravidasvir and sofosbuvir as part of routine clinical practice.

Patients who have initiated antiviral therapy with ravidasvir and sofosbuvir, meet the inclusion criteria, and have signed informed consent for the use of their data in scientific research will be enrolled in the study. Patients will be followed in the clinic in accordance with routine medical practice during the course of ravidasvir and sofosbuvir antiviral therapy.

After 8 weeks of therapy, the rate of viral eradication in peripheral blood will be determined. Patients who achieve a virological response will continue to be followed to assess the maintenance of virological response at 4 and 12 weeks after completion of antiviral therapy.

ELIGIBILITY:
Inclusion Criteria:

* Patient informed consent for the collection and use of data in scientific research.
* Diagnosed chronic hepatitis C (genotype 3).
* Fibrosis stage F0-F2 according to METAVIR, confirmed by liver biopsy or liver elastography (results of performed studies must be no older than 3 months at the start of antiviral therapy).
* Signed informed consent.
* Age ≥18 years.
* Antiviral therapy with ravidasvir and sofosbuvir initiated as part of routine clinical practice.

Exclusion Criteria:

* Significant concomitant liver diseases considered relevant by the investigator (hepatitis B, hemochromatosis, autoimmune hepatitis, primary biliary cholangitis, primary sclerosing cholangitis, hepatocellular carcinoma).
* Presence of other active viral infections (e.g., hepatitis B, HIV).
* If the patient has received other antiviral treatment for hepatitis C within the last 6 months.
* Pregnancy or breastfeeding.
* Alcohol or drug dependence that may interfere with adherence to the treatment regimen.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with chronic hepatitis C virus infection genotype 3 with fibrosis stage F0-F2 were selected for this non-interventional study. These patients represent an important group with a high probability of successful therapy response and relatively low risk of complications, making them ideal candidates for studying the efficacy and safety of a short-term treatment regimen with ravidasvir and sofosbuvir. A similar patient population showed a high rate of sustained virological response (93.42%) in the EASE clinical trial (NCT05757700) with an 8-week therapy regimen. Despite the presence of significant data on treatment of chronic hepatitis C overall, detailed descriptions of disease epidemiology depending on virus genotype, fibrosis stage, and treatment efficacy in patients at early disease stages in real clinical practice are limited.
Sampling Method: Non-Probability Sample
Enrollment: 30 (Actual)
Dates: Start 2025-09-17 (Actual); Primary Completion 2026-02-02 (Estimated); Study Completion 2026-02-02 (Estimated)

PRIMARY OUTCOMES:
Evaluation of the rate of achieving sustained virological response (SVR12) | 20 weeks after enrollment to the study (8 weeks of antiviral treatment + 12 week of post-treatment follow up)
  Absence of detectable hepatitis C virus (HCV) RNA in a patient's blood 12 weeks after completing antiviral treatment

SECONDARY OUTCOMES:
Evaluation of the rate of achieving aviremia 4 weeks after completion of antiviral therapy (SVR-4) | 12 weeks after enrollment (8 weeks of antiviral treatment + 4 weeks of post-treatment follow up)
  The absence of detectable hepatitis C virus (HCV) RNA in a patient's blood 4 weeks after completing antiviral treatment
Assessment of the dynamics of viral load changes during treatment | At Week 4 after enrollment (therapy initiation), at Week 8 after enrollment (end of antiviral treatment), at Week 12 and Week 20 after enrollment (post-treatment follow up).
  The amount of hepatitis C virus RNA present in a milliliter of a patient's blood (IU/mL).
Assessment of the safety and tolerability of therapy. | 20 weeks after enrollment (8 weeks of antiviral therapy and 12 weeks of post-treatment follow up)
  The frequency and nature of side effects associated with the combination of ravidasvir and sofosbuvir.

CONTACTS AND LOCATIONS:
Overall Officials: Pavel Bogomolov, Prof., PhD, MD, Principal Investigator — Center of target therapy
Locations (1):
- Center of Target Therapy LLC., Moscow, Russia

IPD SHARING:
Plan to Share IPD: No